CLINICAL TRIAL: NCT00650260
Title: Intraoperative Warming : Comparison of Performance of the Dynatherm Medical vitalHEAT™ Temperature Management System (vH2) and the Arizant Bair Hugger System
Brief Title: Intraoperative Warming Comparison of Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Dynatherm Medical Inc. (Industry)
Responsible Party: Principal Investigator, Enrico Camporesi, Emeritus Professor of Surgery / Anesthesiology, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 106411c; TGH 100; USF 6176-P67639
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-09

CONDITIONS: Hypothermia
Keywords: intraoperative warming; anesthesia; hypothermia; body temperature
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vH2 System Group (Experimental): The vital heat vH2 system consists of a Control Unit containing the heating system and the vacuum generation pump which connects via an umbilical containing the fluid and vacuum tubing to the Warming Sleeve. The Control Unit also contains the user interface and alarm management systems. The disposable Warming Sleeve consists of a manifold attached to the warming pads and a polyurethane pouch (Vacuum Sleeve) that are placed over the patient's hand and forearm and secured with tape. The Warming Sleeve manifold contains connectors for the fluid and vacuum tubing contained in the umbilical. The vital heat vH2 System will be used for patient warming during these surgical procedures. Monitoring of core temperature via esophageal probe will be done for the purpose of data collection.
  Interventions: Device: Dynatherm Medical vitalHEAT Temperature Management System vH2
- Control Group (Active Comparator): The Bair Hugger system is the current standard of care at Tampa General Hospital. It consists of a Temperature Management Unit that contains the heating element, the air circulating motor and the temperature control mechanisms. This unit connects via a hose to the operating room blankets. The Bair Hugger technology relies on heated air convection. Warm air is circulated evenly through the air space in the specially designed blanket, warming the skin surface as well as any insulating blankets placed over the Bair Hugger blanket. The Bair Hugger System is the site's current approach to patient warming during these surgical procedures. Monitoring of core temperature via esophageal probe will be done for the purpose of data collection.
  Interventions: Device: Bair Hugger™ (Arizant Healthcare, Eden Prairie, MN)

INTERVENTIONS:
Device: Dynatherm Medical vitalHEAT Temperature Management System vH2 — The vH2 system consists of a Control Unit containing the heating system and the vacuum generation pump which connects via an umbilical containing the fluid and vacuum tubing to the Warming Sleeve. The Control Unit also contains the user interface and alarm management systems. The disposable Warming Sleeve consists of a manifold attached to the warming pads and a polyurethane pouch (Vacuum Sleeve) that are placed over the patient's hand and forearm and secured with tape. The Warming Sleeve manifold contains connectors for the fluid and vacuum tubing contained in the umbilical.
  Other Names: Part number VH-200
  Arms: vH2 System Group
Device: Bair Hugger™ (Arizant Healthcare, Eden Prairie, MN) — The Bair Hugger system is the current standard of care at Tampa General Hospital. It consists of a Temperature Management Unit that contains the heating element, the air circulating motor and the temperature control mechanisms. This unit connects via a hose to the operating room blankets. The Bair Hugger technology relies on heated air convection. Warm air is circulated evenly through the air space in the specially designed blanket, warming the skin surface as well as any insulating blankets placed over the Bair Hugger blanket.
  Other Names: Model 522
  Arms: Control Group

SUMMARY:
Hypothermia is a common and serious complication during anesthesia and surgery. Anesthetic-induced hypothermia results from the inhibition of thermoregulatory control and exposure to cold operating room environment.

Various warming methods, such as warm blankets, forced-air warmers and circulating water mattresses, are currently used to prevent and treat mild perioperative hypothermia. All are cutaneous approaches that rely on heating the peripheral tissues in order to increase the thermal core temperature. Application of cutaneous warming system blankets/pads are limited by location/extent of operative site; for example, in certain procedures such as laparatomies, reconstructive plastic surgery or orthopedic surgery, only a limited amount of skin surface is available for warming application. The Dynatherm vitalHEAT technology takes advantage of the body's natural thermoregulatory system to channel thermal energy to the body's core non-invasively at a rapid rate. The vital heat (vH2) system is designed to treat hypothermia during the peri-operative period through a combination of localized heat and vacuum application to one hand & forearm; this application 1) opens the arteriovenous anastamoses located in the palm of the hand and 2) conductively warms the extremity thus effectively warming the blood flow to the body's core. The vital heat vH2 system is a portable and compact warming device which provides a non-invasive approach to warming patients during surgery.

The primary objective of this study is to determine if the Dynatherm Medical vitalHEAT (vH2) Temperature Management System is as effective as the forced-air warming Bair Hugger™ (Arizant Healthcare, Eden Prairie, MN) for maintenance of intraoperative body temperature in patients undergoing abdominal surgery under general anesthesia. The critical endpoints to be evaluated in making this determination are 1) % of subjects with an average intraoperative esophageal temperature of ≥ 36º C and 2) % of subjects with an initial post anesthesia care unit sublingual temperature of ≥ 36º C. Secondary objectives include 1) comparison of the core body temperatures @ 60 minutes post anesthesia induction, 2) comparison of temperature trends during surgery and 3) comparison of the subjects' post anesthesia care unit temperature trends and hypothermic symptoms such as shivering.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective open abdominal surgical procedures with an expected duration of 2 to 4 hours and requiring general anesthesia
* American Society of Anesthesiologists(ASA) physical status I-III
* Patient age: > 18 years and <80 years

Exclusion Criteria:

* Patient age: < 18 years and >80 years
* Patients with break in skin integrity on the extremity selected as the application site
* Patients with history of upper extremity peripheral vascular disease
* Patients with history of allergic skin conditions of the upper extremities
* Patients with history of bleeding disorders/coagulopathy
* Patient with history of malignant hyperthermia
* Patients who are pregnant
* Patient unwilling or unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico M Camporesi, M.D., Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

REFERENCES:
- [Background] Insler SR, Sessler DI. Perioperative thermoregulation and temperature monitoring. Anesthesiol Clin. 2006 Dec;24(4):823-37. doi: 10.1016/j.atc.2006.09.001. PMID 17342966
- [Background] Sessler DI. Perioperative heat balance. Anesthesiology. 2000 Feb;92(2):578-96. doi: 10.1097/00000542-200002000-00042. PMID 10691247
- [Background] Taguchi A, Ratnaraj J, Kabon B, Sharma N, Lenhardt R, Sessler DI, Kurz A. Effects of a circulating-water garment and forced-air warming on body heat content and core temperature. Anesthesiology. 2004 May;100(5):1058-64. doi: 10.1097/00000542-200405000-00005. PMID 15114200
- [Background] Giesbrecht GG, Ducharme MB, McGuire JP. Comparison of forced-air patient warming systems for perioperative use. Anesthesiology. 1994 Mar;80(3):671-9. doi: 10.1097/00000542-199403000-00026. PMID 8141463

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited as they arrived for a scheduled surgical procedure at Tampa General Hospital. Potential subjects were addressed in a private pre-operative room. The investigators or study designee evaluated the patients for the study by reviewing the inclusion and exclusion criteria.
Groups:
- vH2 System Group: The vH2 system consists of a Control Unit containing the heating system and the vacuum generation pump which connects via an umbilical containing the fluid and vacuum tubing to the Warming Sleeve. The Control Unit also contains the user interface and alarm management systems. The disposable Warming Sleeve consists of a manifold attached to the warming pads and a polyurethane pouch (Vacuum Sleeve) that are placed over the patient's hand and forearm and secured with tape. The Warming Sleeve manifold contains connectors for the fluid and vacuum tubing contained in the umbilical. The vH2 System will be used for patient warming during these surgical procedures. Monitoring of core temperature via esophageal probe will be done for the purpose of data collection.
- Control Group: The Bair Hugger system is the current standard of care at TGH. It consists of a Temperature Management Unit that contains the heating element, the air circulating motor and the temperature control mechanisms. This unit connects via a hose to the operating room blankets. The Bair Hugger technology relies on heated air convection. Warm air is circulated evenly through the air space in the specially designed blanket, warming the skin surface as well as any insulating blankets placed over the Bair Hugger blanket. The Bair Hugger System is the site's current approach to patient warming during these surgical procedures. Monitoring of core temperature via esophageal probe will be done for the purpose of data collection.
Period: Overall Study
Arm/Group | vH2 System Group | Control Group
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | vH2 System Group | Control Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 32
  >=65 years | 4 | 6 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 51.1 (18.3) | 46.5 (14) | 48.7 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With an Average Intraoperative Temperature Greater Than or Equal to 36 Celcius
Time Frame: Intraoperative Period
Measure: Number; unit: percentage of participants
Arm/Group | vH2 System Group | Control Group
Number analyzed (Participants) | 21 | 21
percentage of participants | 56 | 90
Statistical Analysis 1: Comparison: vH2 System Group vs Control Group; Test type: Superiority or Other; p = 0.027, Fisher Exact

2. Secondary Outcome: Comparison of the Core Body Temperatures at 60 Minutes Post Anesthesia Induction,as Assessed by Esophageal Probe.
Description: Average core body temperature measured with an esophageal probe at 60 minutes post-induction
Time Frame: 60 minutes post anesthesia induction
Measure: Mean (Standard Deviation); unit: degrees celcius
Arm/Group | vH2 System Group | Control Group
Number analyzed (Participants) | 21 | 21
degrees celcius | 36.4 (0.4) | 36.1 (0.5)
Statistical Analysis 1: Comparison: vH2 System Group vs Control Group; Test type: Superiority or Other; p = 0.078, t-test, 1 sided

3. Secondary Outcome: Average Intraoperative Esophageal Temperature
Description: Average esophageal temperature for the first 70 minutes of surgery following induction of anesthesia.
Time Frame: Intraoperative 0-70 minutes
Measure: Mean (Full Range); unit: Degrees Celcius
Arm/Group | vH2 System Group | Control Group
Number analyzed (Participants) | 21 | 21
Degrees Celcius | 36.3 [35 to 37] | 36.0 [35.1 to 38]

4. Secondary Outcome: Median Post Anesthesia Care Unit Sublingual Temperature
Time Frame: Upon arrival to the post anesthesia care unit
Measure: Median (Full Range); unit: Degrees Celcius
Arm/Group | vH2 System Group | Control Group
Number analyzed (Participants) | 21 | 21
Degrees Celcius | 36.4 [35.9 to 37.4] | 36.6 [36.2 to 37.1]

5. Primary Outcome: Percent of Subjects With an Initial PACU Sublingual Temperature of ≥ 36º C.
Time Frame: Temp taken just prior to surgery
Population: Per protocol, sample size calculations indicate that a total sample size of 42 patients will be necessary to evaluate the primary outcome at an adjusted alpha = 0.05 with 80% power.
Measure: Number; unit: Percentage of participants
Arm/Group | vH2 System Group | Control Group
Number analyzed (Participants) | 21 | 21
Percentage of participants | 95 | 100
Statistical Analysis 1: Comparison: vH2 System Group vs Control Group; Test type: Superiority or Other; p = 1.0, Fisher Exact

6. Primary Outcome: Percentage of Patients With a Post Operative Sublingual Temperature Above 36 Degrees Celcius
Description: Percent of subjects with an initial post anesthesia care unit sublingual temperature of ≥ 36º C
Time Frame: Upon entry to the post anesthesia care unit
Measure: Number; unit: Percentage of participants
Arm/Group | vH2 System Group | Control Group
Number analyzed (Participants) | 21 | 21
Percentage of participants | 95 | 100

ADVERSE EVENTS:
Description: Total number of participants at risk
Arm/Group | vH2 System Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No